CLINICAL TRIAL: NCT00879060
Title: Clinical and Therapeutic Implications of Fibrosis in Hypertrophic Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23HL086745-01A1 (NIH)
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Myocardial Fibrosis; Hypertrophic Cardiomyopathy
Keywords: Fibrosis; Hypertrophic cardiomyopathy; MRI; Myocardial Fibrosis; Spironolactone
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Fibrosis | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spironolactone (Experimental): Experimental group includes individuals diagnosed with HCM between the ages of 18-55 (up to 50 for men). At time of randomization subjects randomized to experimental group will be initiated on 25mg of spironolactone. If at week 4, serum potassium is <5.5 mmol/L and serum creatinine-baseline creatinine is <0.5 mg/dl, the study drug will be increased to the target dose of 50mg once daily.
  Interventions: Drug: Spironolactone
- Placebo Control (Placebo Comparator): Placebo group includes individuals diagnosed with HCM between the ages of 18-55 (up to 50 for men). At time of randomization subjects randomized to placebo group will be initiated on an inactive placebo pill.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — spironolactone 50mg daily
  Other Names: Aldactone
  Arms: Spironolactone
Drug: Placebo — inactive placebo pill daily
  Arms: Placebo Control

SUMMARY:
Hypertrophic Cardiomyopathy (HCM) is the most common genetic cardiomyopathy and remains the leading cause of sudden cardiac death in young people and an important cause of heart failure symptoms and death at any age. In HCM, pathological remodeling of the left ventricle involving myocardial fibrosis is likely a major contributor to cardiac dysfunction and also a nidus for the generation of ventricular arrhythmias. Serum markers of collagen turnover have been shown to reliably reflect the magnitude of myocardial fibrosis in a variety of cardiovascular diseases. In addition, aldosterone antagonist drugs have been shown to decrease fibrous tissue formation in the myocardium in certain pathologic cardiovascular states in which aldosterone production is increased. In HCM, aldosterone production is up-regulated and has been implicated in the formation of myocardial fibrosis.

Therefore, the specific aims of this proposal are to:

1. assess serum markers of collagen turnover at baseline and correlate these findings with a variety of clinical and morphologic disease parameters
2. examine the effects of a 12-month treatment with the aldosterone antagonist spironolactone on magnitude of fibrosis as measured by serum markers of collagen turnover as well as changes in clinical and morphologic disease parameters.
3. explore the effects of a 12-month treatment with aldosterone antagonist spironolactone on heart failure status, diastolic function, arrhythmic burden, and total LV mass and quantity of fibrosis by CMR.

The results of this proposal will offer important insights into the clinical significance of myocardial fibrosis in this primary genetic cardiomyopathy. The demonstration that spironolactone decreases fibrosis and improves clinical course would provide the rational for a larger multicenter clinical trial evaluating this novel therapy for improving clinical outcome in patients with HCM.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is the most common inherited cardiac disease in the general population. Myocardial fibrosis has become a prominent and clinically relevant pathophysiologic component of this complex genetic disease, related to the risk for both sudden death and heart failure. For example, left ventricular replacement fibrosis and scarring has been implicated in triggering life threatening ventricular tachycardia/fibrillation and most recently has become a novel risk marker for sudden death, based on in vivo demonstration of extensive late gadolinium enhancement (LGE) with cardiovascular magnetic resonance (CMR). Extensive LGE identifies patients who benefit from primary prevention of sudden death with the implantable cardioverter-defibrillators (ICD), or who evolve to the end-stage of this disease with systolic dysfunction and consideration for heart transplant.

The mineralocorticoid aldosterone has been shown to be a mediator of myocardial fibrosis, and blockade with spironolactone normalizes collagen content in HCM murine models. In addition, aldosterone antagonists have favorable clinical effects in patients with a variety of diseases associated with myocardial scarring such as congestive heart failure, systemic hypertension, and atherosclerotic coronary artery disease. However, it is uncertain whether spironolactone would have similar effects on the clinical and phenotypic expression of a genetic disease such as HCM. Therefore, we investigated whether mineralocorticoid receptor blockade with spironolactone would reduce measures reflecting myocardial fibrosis, producing favorable LV remodeling and ultimately leading to positive clinical effects for patients with HCM.

The general aim of this study is to explore the role of fibrosis in HCM by testing the hypothesis that: the presence of magnitude of myocardial fibrosis bears clinical relevance for patients with HCM, and that mineralocorticoid receptor blockade will reduce myocardial fibrosis and thereby alter the natural history of the disease.

Experimental design: prospective, randomized, double-blind, placebo-controlled trial in a consecutive HCM population at a single clinical center (Tufts Medical Center HCM Institution).

Study procedures: HCM patients were recruited from Tufts Medical Center HCM Institution population from November 2007 to June 2009. Enrolled patients were randomized into two arms; treatment arm received 25mg at the start of study and then increased to target dose of 50mg if serum potassium was <5.5mmol/L and serum creatinine-baseline creatinine was <0.5mg/dl. This arm was then followed for 12 months. The control arm of the study received 25mg of placebo over 12 months. There was an additional control arm of age and gender-matched controls without HCM in the control arm to evaluate the serum markers of collagen turnover at baseline. These controls had a one time blood draw of 15mL (3 teaspoons) to assess serum biomarkers of interest and were not be followed for 12 months.

Specific outcome measures:

Primary Outcome: examine the effects of a 12-month treatment with the aldosterone antagonist spironolactone on magnitude of fibrosis as measured by serum markers of collagen turnover as well as changes in clinical and morphologic disease parameters.

Secondary Outcomes: explore the effects of a 12-month treatment with aldosterone antagonist spironolactone on heart failure status, diastolic function, arrhythmic burden, and total LV mass and quantity of fibrosis by CMR.

Secondary Outcome: assess serum markers of collagen turnover at baseline and correlate these findings with a variety of clinical and morphologic disease parameters

ELIGIBILITY:
Inclusion Criteria:

1. Hypertrophic cardiomyopathy
2. Able to swallow pills
3. No prior septal reduction therapy
4. Negative serum or hCG pregnancy test

Exclusion Criteria:

1. Unable or unwilling to perform treadmill cardiopulmonary exercise test
2. Prior surgical myectomy or alcohol septal ablation
3. Known or suspected infiltrative or glycogen storage disease
4. Significant coronary artery disease, defined as atherosclerotic coronary artery narrowing >70% of the luminal diameter by coronary angiography
5. Severe obstructive pulmonary disease, defined as forced expiratory volume in 1 second (FEV1) <50% of predicted.
6. Prior intolerance or adverse reaction to aldosterone receptor antagonist.
7. History of hyper or hypoaldosteronism
8. Baseline serum potassium >5.0 mmol/L.
9. Calculated creatinine clearance <30 ml/min using Cockcroft-Gault formula.
10. Pregnant or breast feeding
11. Poorly controlled systemic hypertension, defined as systolic blood pressure ≥150 mmHg or diastolic pressure ≥100 mmHg, during 2 clinic visits.
12. Known conditions associated with elevated serum concentrations of PIIINP (e.g., chronic liver disease, diabetes mellitus, tumors, pulmonary fibrosis, bone and rheumatoid diseases, extensive wounds) or PINP (e.g., alcoholic liver disease, metabolic bone disease, thyroid disorders), including recent trauma (≤2 weeks) or surgery (≤6 months)
13. Taking drugs known to directly influence collagen metabolism including, amiodorone, ACE or angiotensin II inhibitors, aldosterone antagonists, statins, glucocorticoids and estrogens
14. Patients with ICDs/pacemakers will be recruited in the study, but will be excluded from the CMR component.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Maron, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maron BJ, Ommen SR, Semsarian C, Spirito P, Olivotto I, Maron MS. Hypertrophic cardiomyopathy: present and future, with translation into contemporary cardiovascular medicine. J Am Coll Cardiol. 2014 Jul 8;64(1):83-99. doi: 10.1016/j.jacc.2014.05.003. PMID 24998133
- [Background] Chan RH, Maron BJ, Olivotto I, Pencina MJ, Assenza GE, Haas T, Lesser JR, Gruner C, Crean AM, Rakowski H, Udelson JE, Rowin E, Lombardi M, Cecchi F, Tomberli B, Spirito P, Formisano F, Biagini E, Rapezzi C, De Cecco CN, Autore C, Cook EF, Hong SN, Gibson CM, Manning WJ, Appelbaum E, Maron MS. Prognostic value of quantitative contrast-enhanced cardiovascular magnetic resonance for the evaluation of sudden death risk in patients with hypertrophic cardiomyopathy. Circulation. 2014 Aug 5;130(6):484-95. doi: 10.1161/CIRCULATIONAHA.113.007094. PMID 25092278
- [Background] Weng Z, Yao J, Chan RH, He J, Yang X, Zhou Y, He Y. Prognostic Value of LGE-CMR in HCM: A Meta-Analysis. JACC Cardiovasc Imaging. 2016 Dec;9(12):1392-1402. doi: 10.1016/j.jcmg.2016.02.031. Epub 2016 Jul 20. PMID 27450876
- [Background] Lim DS, Lutucuta S, Bachireddy P, Youker K, Evans A, Entman M, Roberts R, Marian AJ. Angiotensin II blockade reverses myocardial fibrosis in a transgenic mouse model of human hypertrophic cardiomyopathy. Circulation. 2001 Feb 13;103(6):789-91. doi: 10.1161/01.cir.103.6.789. PMID 11171784
- [Background] Tsybouleva N, Zhang L, Chen S, Patel R, Lutucuta S, Nemoto S, DeFreitas G, Entman M, Carabello BA, Roberts R, Marian AJ. Aldosterone, through novel signaling proteins, is a fundamental molecular bridge between the genetic defect and the cardiac phenotype of hypertrophic cardiomyopathy. Circulation. 2004 Mar 16;109(10):1284-91. doi: 10.1161/01.CIR.0000121426.43044.2B. Epub 2004 Mar 1. PMID 14993121
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Background] Pitt B, Reichek N, Willenbrock R, Zannad F, Phillips RA, Roniker B, Kleiman J, Krause S, Burns D, Williams GH. Effects of eplerenone, enalapril, and eplerenone/enalapril in patients with essential hypertension and left ventricular hypertrophy: the 4E-left ventricular hypertrophy study. Circulation. 2003 Oct 14;108(15):1831-8. doi: 10.1161/01.CIR.0000091405.00772.6E. Epub 2003 Sep 29. PMID 14517164
- [Background] Braunwald E, Domanski MJ, Fowler SE, Geller NL, Gersh BJ, Hsia J, Pfeffer MA, Rice MM, Rosenberg YD, Rouleau JL; PEACE Trial Investigators. Angiotensin-converting-enzyme inhibition in stable coronary artery disease. N Engl J Med. 2004 Nov 11;351(20):2058-68. doi: 10.1056/NEJMoa042739. Epub 2004 Nov 7. PMID 15531767
- [Background] Pfeffer MA, Pitt B, McKinlay SM. Spironolactone for heart failure with preserved ejection fraction. N Engl J Med. 2014 Jul 10;371(2):181-2. doi: 10.1056/NEJMc1405715. No abstract available. PMID 25006726
- [Background] Pfeffer MA, Claggett B, Assmann SF, Boineau R, Anand IS, Clausell N, Desai AS, Diaz R, Fleg JL, Gordeev I, Heitner JF, Lewis EF, O'Meara E, Rouleau JL, Probstfield JL, Shaburishvili T, Shah SJ, Solomon SD, Sweitzer NK, McKinlay SM, Pitt B. Regional variation in patients and outcomes in the Treatment of Preserved Cardiac Function Heart Failure With an Aldosterone Antagonist (TOPCAT) trial. Circulation. 2015 Jan 6;131(1):34-42. doi: 10.1161/CIRCULATIONAHA.114.013255. Epub 2014 Nov 18. PMID 25406305
- [Background] Shirani J, Pick R, Roberts WC, Maron BJ. Morphology and significance of the left ventricular collagen network in young patients with hypertrophic cardiomyopathy and sudden cardiac death. J Am Coll Cardiol. 2000 Jan;35(1):36-44. doi: 10.1016/s0735-1097(99)00492-1. PMID 10636256
- [Background] Zannad F, Alla F, Dousset B, Perez A, Pitt B. Limitation of excessive extracellular matrix turnover may contribute to survival benefit of spironolactone therapy in patients with congestive heart failure: insights from the randomized aldactone evaluation study (RALES). Rales Investigators. Circulation. 2000 Nov 28;102(22):2700-6. doi: 10.1161/01.cir.102.22.2700. PMID 11094035
- [Background] Querejeta R, Lopez B, Gonzalez A, Sanchez E, Larman M, Martinez Ubago JL, Diez J. Increased collagen type I synthesis in patients with heart failure of hypertensive origin: relation to myocardial fibrosis. Circulation. 2004 Sep 7;110(10):1263-8. doi: 10.1161/01.CIR.0000140973.60992.9A. Epub 2004 Aug 16. PMID 15313958
- [Derived] Maron MS, Chan RH, Kapur NK, Jaffe IZ, McGraw AP, Kerur R, Maron BJ, Udelson JE. Effect of Spironolactone on Myocardial Fibrosis and Other Clinical Variables in Patients with Hypertrophic Cardiomyopathy. Am J Med. 2018 Jul;131(7):837-841. doi: 10.1016/j.amjmed.2018.02.025. Epub 2018 Mar 28. PMID 29604289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects diagnosed with HCM, between the ages of 18-55 (male or female), who are not pregnant were recruited from the Tufts Medical Center Hypertrophic Cardiomyopathy Center. The last patient completed the study in August of 2012.
Groups:
- Spironolactone: Experimental group includes individuals diagnosed with HCM between the ages of 18-55 (up to 50 for men). At time of randomization subjects randomized to experimental group will be initiated on 25mg of spironolactone. Serum potassium and creatinine levels will be drawn at baseline, weeks 1,4,5 and months 3,6,9, and 12. If at week 4, serum potassium is <5.5 mmol/L and serum creatinine-baseline creatinine is <0.5 mg/dl, the study drug will be increased to the target dose of 50mg once daily for 12 months of follow-up. If a subject experiences an increase in serum potassium or creatinine above these parameters at week 4, the study drug will be decreased in half from current dosage. If on 25mg daily, subject will be instructed to decrease to 25mg every other day. Subjects who experience hyperkalemia or increased creatinine levels on 25mg every other day will have the drug discontinued.
- Placebo Control: Placebo group includes individuals diagnosed with HCM between the ages of 18-55 (up to 50 for men). At time of randomization subjects randomized to experimental group will be initiated on 25mg of placebo.
Period: Overall Study
Arm/Group | Spironolactone | Placebo Control
Started | 26 | 27
Completed | 26 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 53 HCM patients (41 +/- 13 years old, 72% men and 28% female) were randomized 1:1 to receive either 50mg of spironolactone or a placebo pill over a 12 month follow up period.
Groups:
- Placebo: spironolactone: spironolactone 50mg daily
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Placebo | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (13) | 42 (13) | 41 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 20 | 18 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Serum Markers of Collagen Turnover (Micrograms/L) Over a One-year Follow-up Period in the Spironolactone Group Compared to Placebo.
Description: Specific variables of collagen turnover markers that will be evaluated include markers of collagen synthesis (PINP, PIIINP), and marker of collagen degradation (ICTP). A two-sample t-test was used to compare the differences between these collagen turnover markers at baseline and the absolute differences in change from baseline to 12 months of follow-up.
Time Frame: The time points measured were at Baseline and at 12 Months (Follow-Up).
Population: 53 HCM patients (41 +/- 13 years old, 72% male) were randomized; demographic, clinical, and structural variables were well matched at baseline.
Measure: Mean (Standard Deviation); unit: micrograms/L
Groups:
- Placebo Control: Placebo group includes individuals diagnosed with HCM between the ages of 18-55 (up to 50 for men). At time of randomization subjects randomized to placebo group will be initiated on 25mg of placebo.
  Placebo: placebo 25mg daily
Arm/Group | Spironolactone | Placebo Control
Number analyzed (Participants) | 26 | 27
micrograms/L
  Baseline (PINP) | 2.1 (1.0) | 2.1 (1.2)
  12 Months (PINP) | 0.7 (12) | 0.6 (1.3)
  Baseline (PIIINP) | 4.7 (2.0) | 4.5 (2.5)
  12 Months (PIIINP) | 2.0 (0.80) | 1.6 (0.80)
  Baseline (ICTP) | 2.2 (1.4) | 2.5 (1.4)
  12 Months (ICTP) | 2.7 (1.4) | -2.3 (1.4)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare continuous variable PINP (serum marker of collagen formation/degradation) between spironolactone treated and placebo groups at baseline; Test type: Other; p = 1.0, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Mean Difference (Final Values) = 0.0
Statistical Analysis 2: Comparison: Placebo Control; A two-sample T-test was used to compare continuous variable PIIINP (serum marker of collagen formation/degradation) between spironolactone treated and placebo groups at baseline; Test type: Other; p = 0.8, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Mean Difference (Final Values) = 0.2
Statistical Analysis 3: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare continuous variable ICTP (serum marker of collagen formation/degradation) between spironolactone treated and placebo groups at baseline; Test type: Other; p = 0.3, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05.aseline; Mean Difference (Final Values) = 0.3
Statistical Analysis 4: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare the absolute differences in change from baseline to 12 months in continuous variable PINP (serum marker of collagen formation/degradation) between spironolactone treated and placebo groups; Test type: Other; p = 1.0, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Absolute difference = 0.0

2. Secondary Outcome: Measure of Functional Capacity: Peak Oxygen Consumption With Exercise
Description: This data was collected at baseline, prior to drug administration, and again at 12-months of follow-up to determine if spironolactone improves a subject's functional capacity during exercise (peak oxygen consumption levels/peak VO2). Peak VO2 levels were measured in ml/kg/min.
Time Frame: The time points measured were at Baseline and at 12 Months (Follow-Up).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Spironolactone | Placebo Control
Number analyzed (Participants) | 26 | 27
ml/kg/min
  Peak VO2 (Baseline) | 30 (7) | 28 (7)
  Peak VO2 (12-Month Follow-Up) | 29 (8) | 29 (6)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare the absolute differences in change from baseline to 12 months in continuous variable peak oxygen consumption with exercise (peak VO2) between spironolactone treated and placebo groups; Test type: Other; p = 0.7, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Absolute difference = 1.2

3. Secondary Outcome: Measure of Heart Failure Symptoms According to the New York Heart Association Functional Class
Description: This data was collected at baseline, prior to drug administration, and again at 12-months of follow-up to assess heart failure symptoms according to the New York Heart Association (NYHA) functional class, which is an estimate of a patients functional ability. The NYHA functional classes include: Class I (no limitation of physical activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity), and Class IV (unable to carry out any physical acitivity without discomfort).
Time Frame: Time points were measured at Baseline and again at 12 months (follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spironolactone | Placebo Control
Number analyzed (Participants) | 26 | 27
score on a scale
  NYHA Class (Baseline) | 1.6 (0.7) | 1.5 (0.6)
  NYHA Class (12-Month Follow Up) | 1.7 (0.8) | 1.6 (0.7)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare the absolute differences in change from baseline to 12 months in continuous variable New York Heart Association (NYHA) Functional Class between spironolactone treated and placebo groups; Test type: Other; p = 0.8, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Absolute difference = 0.0

4. Secondary Outcome: Measure of Indices of Diastolic Function by Tissue Doppler Echocardiography (Septal E/e')
Description: This data was collected at baseline, prior to drug administration, and again at 12-months of follow-up to measure indices of diastolic function by Tissue Doppler Echocardiography using the Septal E/e' ratio.
Time Frame: The time points measured were at Baseline and at 12 Months (Follow-Up).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Spironolactone | Placebo Control
Number analyzed (Participants) | 26 | 27
Ratio
  Diastolic Function (Baseline) | 14 (4) | 15 (7)
  Diastolic Function (12-month Follow-Up) | 13 (6) | 13 (4)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare the absolute differences in change from baseline to 12 months in continuous variable Septal E/e' between spironolactone treated and placebo groups; Test type: Other; p = 1.0, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Absolute difference = 1.4

5. Secondary Outcome: Assessment of Cardiac Mass and Fibrosis by Cardiac Magnetic Resonance Imaging (CMR) - Percentage of Left Ventricular Mass (%LV)
Description: CMR will be utilized as it has superior reproducibility (as compared to 2-D echocardiography). Late Gadolinium Enhancement (LGE) Assessment of myocardial fibrosis by CMR will be expressed as a percentage of left ventricular mass (%LV), maximum left ventricular wall thickness (in mm), left ventricular end-diastolic cavity size (in mm/m^2), and left atrial dimension (in mm).
Time Frame: The time points measured were at Baseline and at 12 Months (Follow-Up).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Total LV Mass
Arm/Group | Spironolactone | Placebo Control
Number analyzed (Participants) | 26 | 27
Percentage of Total LV Mass
  LGE Assessment of Myocardial Fibrosis (Baseline) | 1.1 (2.5) | 2.5 (3.3)
  LGE Assessment of Myocardial Fibrosis (12-Month Follow-Up) | 1.8 (2.9) | 2.8 (4.1)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare the absolute differences in change from baseline to 12 months in continuous variable percentage of left ventricular mass (%LV) between spironolactone treated and placebo groups; Test type: Other; p = 0.7, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Absolute difference = 0.2

6. Secondary Outcome: Assessment of Cardiac Mass and Fibrosis by Cardiac Magnetic Resonance Imaging (CMR) - Maximum Left Ventricular Wall Thickness (in mm)
Description: as for outcome 5
Time Frame: The time points measured were at Baseline and at 12 Months (Follow-Up).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Spironolactone | Placebo Control
Number analyzed (Participants) | 26 | 27
millimeters
  Maximum Left Ventricular Wall Thickness (Baseline) | 22 (7) | 21 (6)
  Maximum Left Ventricular Wall Thickness (12-Month Follow-Up) | 22 (6) | 19 (3)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare the absolute differences in change from baseline to 12 months in continuous variable maximum left ventricular wall thickness (Max LV) between spironolactone treated and placebo groups; Test type: Other; p = 0.4, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Absolute difference = 0.9

7. Secondary Outcome: Assessment of Cardiac Mass and Fibrosis by Cardiac Magnetic Resonance Imaging (CMR) - Left Ventricular End-Diastolic (LVED) Cavity Size (in mm/m^2)
Description: CMR will be utilized as it has superior reproducibility (as compared to 2-D echocardiography). Late Gadolinium Enhancement (LGE) Assessment of myocardial fibrosis by CMR will be expressed as a percentage of left ventricular mass (%LV), maximum left ventricular wall thickness (in mm), left ventricular end-diastolic (LVED) cavity size (in mm/m^2), and left atrial dimension (in mm).
Time Frame: The time points measured were at Baseline and at 12 Months (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/m^2
Arm/Group | Spironolactone | Placebo Control
Number analyzed (Participants) | 26 | 27
mm/m^2
  LVED Cavity Size (Baseline) | 133 (26) | 145 (46)
  LVED Cavity Size (12-Month Follow-Up) | 129 (29) | 146 (44)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare the absolute differences in change from baseline to 12 months in continuous variable left ventricular end-diastolic (LVED) cavity size between spironolactone treated and placebo groups; Test type: Other; p = 0.7, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Absolute difference = 5.7

8. Secondary Outcome: Assessment of Cardiac Mass and Fibrosis by Cardiac Magnetic Resonance Imaging (CMR) - Left Atrial Dimension (in mm)
Description: as for outcome 5
Time Frame: The time points measured were at Baseline and at 12 Months (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Spironolactone | Placebo Control
Number analyzed (Participants) | 26 | 27
millimeters
  Left Atrial Dimension (Baseline) | 40 (6) | 41 (5)
  Left Atrial Dimension (12-Month Follow-Up) | 40 (5) | 40 (6)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo Control; A two-sample T-test was used to compare the absolute differences in change from baseline to 12 months in continuous variable left atrial dimension between spironolactone treated and placebo groups; Test type: Other; p = 0.8, t-test, 2 sided — An a priori threshold for statistical significance was determined at an alpha level of 0.05; Absolute difference = 0.1

ADVERSE EVENTS:
Groups:
- Control Group: A control population of age and gender-matched volunteers recruited from the general medicine outpatient clinic at Tufts Medical Center as well as from Tufts Medical Center employees. Controls will be excluded if any history of heart disease or any risk factors for cardiovascular disease, conditions of physiological or pathological activation of collagen turnover. Control subjects will have a one time blood draw of 16mL (3 teaspoons).
Arm/Group | Spironolactone | Control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

LIMITATIONS AND CAVEATS:
Study population was small in size; duration of drug administration of 1 year too abbreviated to identify clinical/ structural changes in HCM; 50% patients asymptomatic (peak VO2 normal) limit opportunity for improvement with drug intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes